CLINICAL TRIAL: NCT05478681
Title: Home-based tDCS for Behavioral Symptoms in Alzheimer's Disease and Related Dementias (ADRD)
Brief Title: Home-based Transcranial Direct Current Stimulation (tDCS) for Behavioral Symptoms in Alzheimer's Disease and Related Dementias (ADRD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Texas Alzheimer's Research and Care Consortium (Other)
Responsible Party: Principal Investigator, Kendra Anderson, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-22-0296
Record Dates: First submitted 2022-07-25; First posted 2022-07-28 (Actual); Results first posted 2025-10-10 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-09

CONDITIONS: Alzheimer Disease
Keywords: depression; anxiety; irritability; apathy; psychosis; tDCS
MeSH Terms: conditions — Alzheimer Disease; Depression; Anxiety Disorders; Lethargy; Psychotic Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- active tDCS (Experimental): All participants will receive active tDCS with a constant current intensity of 2mA. Anodal tDCS will be applied to the left dorsolateral prefrontal cortex, while cathodal electrode will be positioned on the right dorsolateral prefrontal cortex. Caregivers will help setting up and administering tDCS for participants with AD at home. tDCS will be applied for 30min at an intensity of 2mA, with 30 s ramping up and down.
  Interventions: Device: active tDCS

INTERVENTIONS:
Device: active tDCS — All participants will receive active tDCS with a constant current intensity of 2mA. Anodal tDCS will be applied to the left dorsolateral prefrontal cortex, while cathodal electrode will be positioned on the right dorsolateral prefrontal cortex. Caregivers will help setting up and administering tDCS for participants with AD at home. tDCS will be applied for 30min at an intensity of 2mA, with 30 s ramping up and down.

SUMMARY:
The purpose of this study is to assess acceptability, and safety of providing tDCS to ADRD patients with behavioral symptoms and to assess the efficacy of tDCS for ADRD-related symptoms, mainly behavioral symptoms.

ELIGIBILITY:
Inclusion Criteria:

* have ADRD and clinically-meaningful behavioral symptoms
* have a caregiver willing to participate in the study
* can speak and read English
* have stable doses of medications for at least one month

Exclusion Criteria:

* any unstable concurrent medical conditions
* history of brain surgery
* seizure
* intracranial metal implantation
* current alcohol/substance use disorder

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2023-04-17 (Actual); Primary Completion 2024-02-26 (Actual); Study Completion 2024-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kendra M Anderson, PhD, Principal Investigator — The University of Texas Health Science Center, Houston; Antonio L Teixeira, MD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (2):
- United States (2):
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active tDCS
Started | 3
Completed | 1
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: Only 3 participants were enrolled in this study. Of the 3 participants only 1 completed the study. Based on the low enrollment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Arm/Group | Active tDCS
Number analyzed (Participants) | 0
Age, Categorical
Sex: Female, Male
Ethnicity (NIH/OMB)
Race (NIH/OMB)
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Acceptability of the tDCS Treatment as Assessed by the tDCS Acceptability Questionnaire
Description: The tDCS acceptability questionnaire has a total score from 0 to 100, a higher score indicates higher acceptance of the tDCS treatment.
Time Frame: week 2
Population: as for baseline characteristics
Arm/Group | Active tDCS
Number analyzed (Participants) | 0

2. Primary Outcome: Acceptability of the tDCS Treatment as Assessed by the tDCS Acceptability Questionnaire
Description: as for outcome 1
Time Frame: week 4
Population: as for baseline characteristics
Arm/Group | Active tDCS
Number analyzed (Participants) | 0

3. Primary Outcome: Acceptability of the tDCS Treatment as Assessed by the tDCS Acceptability Questionnaire
Description: as for outcome 1
Time Frame: week 6
Population: as for baseline characteristics
Arm/Group | Active tDCS
Number analyzed (Participants) | 0

4. Primary Outcome: Acceptability of the tDCS Treatment as Assessed by the tDCS Acceptability Questionnaire
Description: as for outcome 1
Time Frame: week 12
Population: as for baseline characteristics
Arm/Group | Active tDCS
Number analyzed (Participants) | 0

5. Primary Outcome: Safety as Assessed by the Side Effects Questionnaire
Description: side effects include itching, burning, headache, fatigue, and dizziness.
Time Frame: week 2
Population: as for baseline characteristics
Arm/Group | Active tDCS
Number analyzed (Participants) | 0

6. Primary Outcome: Safety as Assessed by the Side Effects Questionnaire
Description: side effects include itching, burning, headache, fatigue, and dizziness.
Time Frame: week 4
Population: as for baseline characteristics
Arm/Group | Active tDCS
Number analyzed (Participants) | 0

7. Primary Outcome: Safety as Assessed by the Side Effects Questionnaire
Description: side effects include itching, burning, headache, fatigue, and dizziness.
Time Frame: week 6
Population: as for baseline characteristics
Arm/Group | Active tDCS
Number analyzed (Participants) | 0

8. Secondary Outcome: Dementia-related Behavioral Symptoms as Assessed by the Neuropsychiatric Inventory (NPI-Q) Scale
Description: NPI-Q evaluates 12 discrete neuropsychiatric symptoms considering their severity and the related caregiver distress.
Time Frame: Baseline, week 2, week 4, week 6, week 12
Population: as for baseline characteristics
Arm/Group | Active tDCS
Number analyzed (Participants) | 0

9. Secondary Outcome: Apathy as Assessed by the Brief Dimensional Apathy Scale (b-DAS)
Description: This scale consists of 9 questions each one scored from 0(almost always) to 3(hardly ever), higher scores indicate more apathy
Time Frame: Baseline, Week 6 and Week 12.
Population: as for baseline characteristics
Arm/Group | Active tDCS
Number analyzed (Participants) | 0

10. Secondary Outcome: Depressive Symptoms as Assessed by the Cornell Scale for Depression in Dementia (CSDD)
Description: This questionnaire has 19 questions and each is scored from 0(absent) to 2(severe). A total score greater than 10 indicates probable major depressive episode and a score of greater than 18 indicates definite major depressive episode
Time Frame: Baseline, Week 6 and Week 12.
Population: as for baseline characteristics
Arm/Group | Active tDCS
Number analyzed (Participants) | 0

11. Secondary Outcome: Cognition as Evaluated by the Mini-Mental State Examination (MMSE)
Description: Mini-Mental State Examination (MMSE) includes memory, language, praxis and orientation tasks, yielding a global cognition score ranging 0 to 30, with higher scores indicating better performance.
Time Frame: Baseline, Week 6 and Week 12.
Population: as for baseline characteristics
Arm/Group | Active tDCS
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Only 3 participants were enrolled in this study. Of the 3 participants only 1 completed the study. Based on the low enrollment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Description: Only 3 participants were enrolled in this study. Of the 3 participants only 1 completed the study. Based on the low enrollment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Arm/Group | Active tDCS
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-27): https://cdn.clinicaltrials.gov/large-docs/81/NCT05478681/Prot_SAP_000.pdf